CLINICAL TRIAL: NCT04189536
Title: An SMS Intervention to Improve Adherence to Stimulant Medications in Adults With ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Joseph Biederman, MD, Chief of the Clinical and Research Programs in Pediatric Psychopharmacology and Adult ADHD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-P-001087
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Attention Deficit/Hyperactivity Disorder
Keywords: Attention Deficit/Hyperactivity Disorder; ADHD; SMS Intervention
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMS Intervention (Experimental): All subjects will receive customized text messages twice a day, every day for 9 months that will include reminders to adhere to the individualized medication regimen, reminders to call their clinician for a prescription refill followed by reminders to pick up medication from the pharmacy, and educational reminders about ADHD and its treatment.
  Interventions: Other: SMS Intervention

INTERVENTIONS:
Other: SMS Intervention — Delivery of text messages will use the Rip Road Mobile platform.

SUMMARY:
This study will assess the efficacy of the text messaging (SMS-based) disease management intervention to improve adherence to stimulants in adults with Attention Deficit/Hyperactivity Disorder (ADHD).

Participants in the study will receive customized text messages twice a day, every day, for a duration of 9 months. The text messages will include reminders to adhere to the individualized medication regimen, reminders to call their clinician for a prescription refill followed by reminders to pick up medication from the pharmacy, and educational reminders about ADHD and its treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults 18 to 55 years
* A diagnosis of Diagnostic and Statistical Manual Diploma in Social Medicine (DSM-V) Attention Deficit Hyperactivity Disorder based on clinical assessment
* Is starting stimulant medication or has begun treatment with stimulant medication within six months of study enrollment
* Proficient in English
* Has a cellular phone with text messaging capabilities and is interested in and willing to receive text messages

Exclusion Criteria:

* Serious chronic medical or psychiatric condition that, in the investigator's opinion, puts the subject at risk for taking a stimulant
* Pregnant or nursing females
* Investigator and his/her immediate family
* Unwilling/unable to comply with study procedures

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Estimated)
Dates: Start 2016-09-19 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Adherence to Stimulants | 9 months
  Adherence will be analyzed using the timeliness of stimulant medication prescription renewals over the 9 month period.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No